CLINICAL TRIAL: NCT02835950
Title: Clinical Evaluation of the Therapeutic Intra-Vascular Ultrasound (TIVUS™) System for Pulmonary Artery Denervation (PDN) in Patients With Pulmonary Hypertension - US
Brief Title: TReatment Of Pulmonary HYpertension 1-US Study
Acronym: TROPHY 1-US
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SoniVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNS01-001 USA
Record Dates: First submitted 2016-07-10; First posted 2016-07-18 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Pulmonary Denervation (Experimental): Pulmonary Denervation (PDN) using the TIVUS™ System will be performed in patient suffering from pulmonary arterial hypertension after completion of screening and eligibility phase, The procedure will be performed during right heart catheterisation. Safety and effectiveness of the PDN treatment will be assessed during one year follow up.
  Interventions: Device: Therapeutic Intra-Vascular UltraSound (TIVUS™) System

INTERVENTIONS:
Device: Therapeutic Intra-Vascular UltraSound (TIVUS™) System — The TIVUS™ System generates high intensity, non-focused ultrasonic energy that is delivered through the wall of the pulmonary artery to achieve local nerve deactivation.
  Denervation in the pulmonary arteries (PDN) would be performed during right heart catheterization. The PDN procedure would be attempted in the main, right and left pulmonary arteries, close to the main bifurcation.
  Other Names: TIVUS™

SUMMARY:
The objective of this study is to assess the safety, performance and initial effectiveness of the TIVUS™ System when used for pulmonary artery denervation through subjective and objective change in clinical parameters and haemodynamic evaluation. This is a prospective, multi-center, non-randomized, open-label clinical trail. The study will be conducted in up to 4 centers and will recruit up to 15 patients diagnosed with PAH, functional class III who have stable PAH on a stable drug regimen of two pulmonary arterial hypertension specific medications.

ELIGIBILITY:
Inclusion Criteria:

* Patient with known pulmonary arterial hypertension (PAH), diagnosed as idiopathic PAH, connective tissue disease PAH, Anorexogen induced or Heritable PAH
* PAH diagnosis confirmed by hemodynamic evaluation performed prior to screening and showing all of the following: Mean pulmonary artery pressure (mPAP) ≥25 mmHg at rest; Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤15 mmHg; Pulmonary vascular resistance (PVR) at rest >3 Wood units; Not meeting the criteria for a positive vasodilator response (fall in mPAP ≥ 10 mmHg to ≤ 40 mmHg).
* Patient with a current diagnosis of WHO functional class III
* Patient taking two pulmonary arterial hypertension specific medications other than parenteral prostanoids
* Patient is adhering to a stable drug regimen (i.e., with no changes of dose or medication for a minimum of 3 months prior to enrollment)
* Patient with eGFR levels of ≥ 30 ml/min/1.73m2or serum creatinine levels of ˂ 150µmol/l

Exclusion Criteria:

* Patients who are treated with parenteral prostanoids
* Pregnant women or women planning a pregnancy within 12 months of study enrolment
* Patient with significant co-morbid condition(s) which, at the discretion of the PI, are deemed to prohibit study entry
* Patient with life expectancy of less than a year
* Concurrent enrollment in another device or drug trial except for observational studies (unless specifically approved by the sponsor)
* Patient with pulmonary artery anatomy that precludes treatment
* Patient with moderate to severe pulmonary artery stenosis
* Patient with any pulmonary artery aneurysm
* Patient who has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident in the previous 6 months
* Patient who has implantable cardiac pacemakers, ICDs, neurostimulators, or drug infusion devices
* Patients who are unable to undergo an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Amount of all procedural related adverse event as assessed by the CEC | 1 month
  Procedural related Adverse Events
Amount of treatment related adverse event as assessed by the CEC | 12 month
  All treatment related adverse events
Number of patient with PAH worsening and all cause death events | 12 month
  PAH related adverse events and all cause death

SECONDARY OUTCOMES:
Clinical effectiveness | 6 months
  Changes from baseline of mean pulmonary arterial pressure (mPAP)
Clinical effectiveness | 6 months
  Changes from baseline of pulmonary vascular resistance (PVR)
Clinical effectiveness | 6 months
  Changes from baseline of 6 minute walking distance (6MWD)
Clinical effectiveness | 6 months
  Changes from baseline of quality of life questionaire
Clinical effectiveness | 1, 6 and 12 months
  NT-pro-BNP levels
Clinical efffectivness | 6 months
  Change from baseline in Right Ventricular (RV) function as assesed by MRI
Clinical efffectivness | 6 months
  Change from baseline in Right Ventricular (RV) function as assesed by Echocardiography

OTHER OUTCOMES:
Observational Variables | 12 Months
  Changes from baseline of mean pulmonary arterial pressure (mPAP)
Observational Variables | 12 Months
  Changes from baseline of pulmonary vascular resistance (PVR)
Observational Variables | 12 Months
  Changes from baseline of 6 minute walking distance (6MWD)
Observational Variables | 12 Months
  Changes from baseline of quality of life questionaire
Observational Variables - Long term surveillance | 2, 3, 4 and 5 years
  Clinical change of pulmonary arterial hypertension condition defined by patient survival or cause of mortality
Observational Variables - Long term surveillance | 2, 3, 4 and 5 years
  Clinical change of pulmonary arterial hypertension condition defined by hospitalization due to pulmonary arterial hypertension
Observational Variables - Long term surveillance | 2, 3, 4 and 5 years
  Clinical change of pulmonary arterial hypertension condition defined by any intervention or surgical procedures the patient did
Observational Variables - Long term surveillance | 2, 3, 4 and 5 years
  Clinical change of pulmonary arterial hypertension condition defined by worsening of WHO functional class
Observational Variables - Long term surveillance | 2, 3, 4 and 5 years
  Clinical change of pulmonary arterial hypertension condition defined by escalation of drug therapy
Observational Variables | 12 month
  Echocardiography parameters

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UC San Diego Health, San Diego, California
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University Medical Center/NewYork Presbyterian Hospital, New York, New York
  - UT Southwestren Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No